CLINICAL TRIAL: NCT00722215
Title: The Systemic & Renal Effects of Endothelin Receptor Antagonism in Proteinuric Nephropathy
Brief Title: Endothelin Receptor Antagonism in Proteinuric Nephropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Dr Neeraj Dhaun, The University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2006/WCRC/02; PG/05/91; 06/MRE00/12
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2006-08

CONDITIONS: Chronic Kidney Disease; Proteinuria
Keywords: Endothelin antagonist; Chronic kidney disease; Proteinuria; Cardiovascular disease; Blood pressure; Arterial stiffness; Endothelial function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria; Cardiovascular Diseases | interventions — cyclo(Trp-Asp-Pro-Val-Leu); Sodium Chloride; Nifedipine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo control arm of study
  Interventions: Drug: 0.9 % saline
- 2 (Experimental): BQ-123 arm of study
  Interventions: Drug: BQ-123 (selective endothelin A receptor antagonist)
- 3 (Active Comparator): Nifedipine arm of study
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: BQ-123 (selective endothelin A receptor antagonist) — Single dose of BQ-123 given at a dose of 1000 nmol/min for 15 min intravenously.
  Arms: 2
Drug: 0.9 % saline — Single 15ml 0.9% saline infused for 15 mins as placebo control
  Arms: 1
Drug: Nifedipine — Single dose of nifedipine 10 mg given orally as active control
  Other Names: Adalat
  Arms: 3

SUMMARY:
The number of people with kidney problems is increasing rapidly, related in part to the increasing prevalence of diabetes. Patients with kidney problems tend to have protein leaking into the urine (proteinuria). Both proteinuria and the kidney disease itself are associated with an increased risk of heart disease. Reducing proteinuria is an important treatment goal in people with kidney problems. Endothelin is a chemical produced both by blood vessels and the kidney. Higher than normal levels of endothelin are thought to contribute to progression of kidney disease and proteinuria. By using drugs that block the effects of endothelin ('endothelin receptor antagonists') we can hopefully reduce both of these. The purpose of the study is to ascertain whether endothelin receptor antagonists improve kidney function and reduce proteinuria more so than other commonly used drugs.

DETAILED DESCRIPTION:
Response to ETA Receptor Antagonism/Nifedipine/Placebo Prior to the study visit subjects will be asked to refrain from alcohol for 24 hours. Tea and coffee will not be permitted for at least 12 hours before each visit. Studies will be conducted in a quiet, temperature-controlled room.

On arrival at the Clinical Research Centre on the study day, a brief medical enquiry and examination will confirm the ongoing suitability of the subject for the study. An intravenous cannula will be inserted into the antecubital fossa of each arm. We have developed a basic protocol described fully in our previous studies that allows us to measure systemic haemodynamics by the well validated technique of bioimpedance and renal function by standard para-aminohippurate (PAH; renal blood flow) and inulin (glomerular filtration rate) clearance studies.

Urinary protein excretion will be measured by collecting urine over 30 minute time periods. To ascertain the contribution of renal haemodynamics to any change in protein excretion renal blood flow and glomerular filtration rate will be measured. In addition, blood and urine will also be assayed for sodium, creatinine and osmolality to allow calculation of fractional excretion of sodium and free water clearance.

Systemic haemodynamic monitoring will be performed at 15 minute intervals during drug/placebo administration and at 30 minute intervals outwith these periods.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-70
* Body mass index <35
* Blood pressure <160/110 mmHg
* CKD stage 2-5 as per the K/DOQI classification
* Proteinuria in one of the following categories: 0.3-1.5, >1.5-3.0, and >3.0-6.0 g/24hrs
* Normal serum albumin

Exclusion Criteria:

* Subject is below the age of legal consent, or is mentally or legally incapacitated
* History of multiple and/or severe allergic reactions to drugs (including study drugs), or food
* The subject has donated blood (450 ml) within the last 4 weeks
* Past or present drug or alcohol abuse including intravenous drug abuse at any time
* Participation in another clinical trial within 1 month
* Considered to be at high risk of HIV or hepatitis B
* Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Proteinuria | Acute change in proteinuria over 4 hour period following BQ-123 dosing
Blood pressure | Acute change in blood pressure over 4 hour period following BQ-123 dosing

SECONDARY OUTCOMES:
Arterial stiffness (as measured by pulse wave velocity) | Acute change in arterial stiffness over 4 hour period following BQ-123 dosing
Endothelial function (as measured by flow-mediated dilatation) | Acute change in endothelial function over 4 hour period following BQ-123 dosing

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Dhaun, MBChB, Principal Investigator — University of Edinburgh; David J Webb, MD, Study Director — University of Edinburgh
Locations (1):
- Clinical Research Centre, Western General Hospital, Edinburgh, Scotland, United Kingdom